CLINICAL TRIAL: NCT04057755
Title: Double Blind Placebo-controlled RCT of the Efficacy and Safety of Intramuscular Injections of Botulinum Toxin A as a Treatment for Provoked Vestibulodynia
Brief Title: Botulinum Toxin A as a Treatment for Provoked Vestibulodynia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Nina Bohm-Starke, MD, associte professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016-000375-25
Record Dates: First submitted 2018-03-06; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Vulvodynia
Keywords: botulinum toxin A; treatment
MeSH Terms: conditions — Vulvodynia | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Botulinum toxin A vs placebo (Experimental): 50 Allergan units (diluted in 0,5 ml sterile NaCl) or 0,5 ml of sterile NaCl will be injected in the bulbocavernosus muscle just inside the hymenal ring. The injection with the same substance, dose and volume will be repeated after 3 months.
  Interventions: Drug: botulinum toxin A; Drug: NaCl
- Botulinum toxin A (Active Comparator): 50 Allergan units (diluted in 0,5 ml sterile NaCl) will be injected in the bulbocavernosus muscle just inside the hymenal ring. The injection with the same substance, dose and volume will be repeated after 3 months.
  Interventions: Drug: botulinum toxin A
- NaCl (Placebo Comparator): 0,5 ml of sterile NaCl will be injected in the bulbocavernosus muscle just inside the hymenal ring. The injection with the same substance and volume will be repeated after 3 months.
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: botulinum toxin A
  Other Names: Botox
  Arms: Botulinum toxin A; Botulinum toxin A vs placebo
Drug: NaCl
  Other Names: Saline
  Arms: Botulinum toxin A vs placebo; NaCl

SUMMARY:
Women with provoked vestibulodynia (PVD) suffer from severe dyspareuni and often present a hyperactivity of the pelvic floor muscles (PFM) which maintain the dyspareunia. The rationale for the study is that for women with PVD who don't succeed to restore the function of the PFM by physiotherapy, Botulinum Toxin A (BTA) could be an optional treatment by decreasing the high muscle tonus and thus possibly reduce the coital pain.

Objectives and outcome Women with PVD will be recruited for a double blind RCT of 2 injection of 50 Allergan-units BTA (3 months apart) or placebo in the bulbocavernous muscles (situated adjacent to the lower part of the vagina).

Primary outcome: The reduction of patient self-reported dyspareunia measured by VAS 0 (no pain) to 100 (worst pain imaginable).

Secondary outcome: Pain at tampon insertion measured by VAS 0-100, functional measurement of dyspareunia (see below), the reduction of pelvic floor hyperactivity/tonus, measured with a vaginal manometer, safety aspects and effect duration of BTA, influence on quality of life and psychosexual evaluation.

DETAILED DESCRIPTION:
Rationale Dyspareunia is a common pain problem among women. The prevalence has been estimated to be 10-15%. The most common type of dyspareunia among premenopausal women is provoked vestibulodynia (PVD). PVD is characterized by pain upon touch, pressure and stretch of the vestibular tissue in spite of the absence of other gynecological or dermatological disease [4]. The pain and its associated sexual consequences have a severe negative impact on the quality of life of affected women. Currently the etiology, although still not completely clarified, is considered to be multi-factorial involving biomedical and psychosexual causes. Two sub-categories of PVD has been identified; primary PVD, where pain occurs at the first attempt of vaginal entry (intercourse or tampon use) and secondary PVD, where pain occurs after a period of normal functioning. There is evidence of patho-physiological changes in three interdependent systems; the vestibular tissue, the pelvic floor muscles and the pain regulatory pathways of the central nervous system. Signs of a neurogenic inflammation in the vestibular mucosa, with neural hyperplasia of CGRP and Substance P positive C-fibers have been found. Furthermore, recent evidence supports the importance of a pelvic floor muscle (PFM) dysfunction to the etiology of PVD. Women with PVD have been shown to have elevated resting activity, lower maximal strength and poorer control of the PFM compared to healthy controls. Evidence suggests that this hyperactivity, although possibly originating as a protective defense mechanism provoked by pain, is chronic and thus contributes to maintaining and exacerbating the neurogenic inflammation and pain. A circular model has been suggested in which pain during intercourse and fear of pain may decrease sexual arousal and increase PFM tonus, whereby the PFM hyperactivity might act as an initiator of vestibular sensory changes and inflammation. However there is a lack of longitudinal studies to answer the question whether the PFM dysfunction is antecedent to the pain or a result of the pain.

Gentilcore-Saulnier et al. proposed that superficial and deep layers of the PFM may differ in their involvement in PVD as assessed with EMG external surface electrodes and an intravaginal probe, respectively. They found that women with PVD have significantly higher resting activity in the superficial muscle (bulbocaverneous) in comparison with controls. The difference was not significant for the deep layer (puborectalis, pubococcygeus, ileococcygeus and ischiococcygeus muscles).

The treatment guidelines today recommend a multi-modal treatment including topical anesthetic agents, cognitive behavioral therapy and PFM rehabilitation based on physiotherapy. As a second line treatment injections with botulinum toxin A (BTA) in the bulbocavernous muscles bilaterally has been suggested and to a limited extent tested. The main target for BTA is a transient paretic effect on skeletal muscular fibers and it also blocks the release of neuropeptides and neurotransmitters involved in the neuropathic pain and could therefore have additional effect in the treatment of PVD. Previously published reports on the effects of BTA for PVD are few and the methods of injection (different injection sites, use or non-use of an EMG needle for direction of injection sites) and doses used (20, 35, 100 IU) differ as well as methods of measuring treatment outcome. Only one double blind RCT has been published so far where no additional effect of BTA compared to saline could be detected, however the BTA dose used was low (20 IU) and only one treatment was performed. Using BTA in the PFM seems to be safe and only tenderness at the injection site and mild influenza like symptoms have been reported side effects so far.

Hypothesis Our hypothesis is that two treatments (three months apart) of injections with 50 Allergan-units of BTA in the bulbocavernosus muscles in women with PVD will reduce the hyperactivity in the PFM and thus significantly decrease the pain during intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* PVD defined as significant pain at vestibular contact and vaginal entry
* VAS ≥ 6 at the tampon test or severe pain, preventing intercourse
* Duration of symptoms of ≥ 3 months
* 0-para
* Patients who are willing to participate in the study after it has been explained orally and in writing will be included.

Exclusion Criteria:

* Vulvo-vaginal infection
* Dermatological conditions or other causes to dyspareunia
* Regular medication with analgesics
* Major psychiatric or medical disease
* Known allergy to any components of the active drug (Botox®)
* Medical disease contradictory to treatment with the active drug (Botox®)
* Peripheral motor neurological disease such as myasthenia gravis, amyotrophic lateral sclerosis or Lambert-Eaton syndrome
* Diabetes)
* Pregnancy
* Pelvic floor deficiency with urine and or flatulence incontinence.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change in self-reported dyspareunia last month measured by VAS 0-100 | At baseline up to 6 months
  VAS 0 (no pain) to 100 (worst pain imaginable).

SECONDARY OUTCOMES:
Change in pain at tampon insertion last week, measured by VAS 0-100 | At baseline and up to 12 months
  VAS 0 (no pain) to 100 (worst pain imaginable).
Change in pelvic floor hyperactivity/tonus, | At baseline and up to 12 months
  Measured with a vaginal manometer in mmHg
Safety aspects regarding adverse events of BTA | The complete study, 12 months
  Monitoring possible adverse events
Change in quality of Life (WHOQOL-BREF) | At baseline and up to 12 months
  The validated questionnaires WHO Quality of Life-BREF (WHOQOL-BREF) will be used
Change in quality of Life (EQ5D) | At baseline and up to 12 months
  Health-related quality of life as assessed using the EuroQOL five dimensions
Change in sexual function | At baseline and up to 12 months
  The validated questionnaire Female Sexual Function Index (FSFI) will be used
Change in sexual distress | At baseline and up to 12 months
  The validated questionnaire Female Sexual Distress Scale (FSDS) will be used
Change in level of stress | At baseline and up to 12 months
  The validated questionnaire PSS (Percieved stress scale) will be used
Change in level of anxiety | At baseline and up to 12 months
  A validated questionnaire Adult Anxiety Scale will be used,

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bohm-Starke, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyd Hospital, Dep. of Obstetrics and Gynecology, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No